CLINICAL TRIAL: NCT01616147
Title: LIFT: Lifestyle Interventions For Two (Member of the LIFE Moms Consortium)
Brief Title: LIFT: Lifestyle Interventions For Two
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dympna Gallagher, Professor of Nutritional Medicine at CUMC, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAO0651; 1U01DK094463 (NIH)
Record Dates: First submitted 2012-06-07; First posted 2012-06-11 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Overweight; Pregnancy
Keywords: Intensive Lifestyle Intervention
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Lifestyle Intervention (ILI) (Experimental): Women in the ILI arm will receive intensive counseling during pregnancy and group counseling after delivery regarding behavior, nutrition, and physical activity change. Visits to counselors will occur twice monthly with additional weekly telephone and internet contacts.
  Interventions: Behavioral: Intensive Lifestyle Intervention (ILI)
- Usual Care (Active Comparator): Women in the usual care group will be offered group support classes approximately every 2 months during pregnancy and 3 months after pregnancy.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention (ILI) — Women in the ILI arm will receive intensive counseling during pregnancy and group counseling after delivery regarding behavior, nutrition, and physical activity change. Visits to counselors will occur twice monthly with additional weekly telephone and internet contacts.
  Arms: Intensive Lifestyle Intervention (ILI)
Behavioral: Usual Care — Women in the usual care group will be offered group support classes approximately every 2 months during pregnancy and 3 months after pregnancy.
  Arms: Usual Care

SUMMARY:
This randomized, controlled trial is proposed to study the effect, in a cohort of racially and ethnically diverse group of overweight and obese pregnant women, of an Intensive Lifestyle Intervention (ILI) which utilize cognitive behavioral strategies to help participants achieve and maintain changes in dietary intake and physical activity habits compared to Usual Care (UC) on gestational weight gain (GWG), infant fatness, and mothers' post-delivery weight retention. The hypothesis is that the percent body fat at birth will be significantly less in offspring from ILI mothers than UC mothers.

DETAILED DESCRIPTION:
Overall body weight and weight gain during pregnancy have gone up among all women in the United States. Higher body weight of the mother at the time of the baby's conception and a greater weight gain during pregnancy are both associated with more fat in the infant and later overweight in children. Obesity in children has become a great public health problem. This study will use the new Institute of Medicine Guidelines for weight gain during pregnancy. These Guidelines are based on observations showing that women whose weight gain was within the recommended Guidelines had healthier pregnancies and better pregnancy outcomes than those who did not follow the Guidelines. It is important for researchers to understand whether a lifestyle intervention like LIFT can help women have healthier pregnancies and healthier babies. If the researchers find that a lifestyle intervention positively impacts the mothers and their babies, then the researchers can help other pregnant women have healthier pregnancies and babies as well.

This Study, The Lifestyle Intervention For Two (LIFT) Study, is part of the LIFE Moms consortium, a national project involving seven sites across the US. The purpose of the LIFE Moms consortium is to study different ways in which women who are overweight or obese can manage their body weight during pregnancy, and how this may affect them and their baby's health at birth and through the first year. As part of the LIFE Moms consortium, The LIFT Study will look how controlled weight gain during pregnancy will impact the health of the mother and her child. Researchers at Columbia University are investigating the effect of an intensive lifestyle intervention (i.e. diet and physical activity counseling). The researchers hope to positively impact not only body weight gain during pregnancy, but also positively impact infant body fatness and mother's weight loss after pregnancy. The LIFE Moms researchers are looking at whether too much weight gain in the mother will result in a leaner baby, and less retention of fat by the mother following pregnancy.

This study is a randomized controlled trial to study the effect, in a cohort of racially and ethnically diverse group of overweight and obese pregnant women, of an Intensive Lifestyle Intervention (ILI) compared to Usual Care (UC) on gestational weight gain (GWG), infant fatness, and mothers' post-delivery weight retention. Women in the ILI arm will receive intensive counseling during pregnancy and group counseling after delivery regarding behavior, nutrition, and physical activity change. Visits to counselors will occur semi-monthly and additional telephone and internet contacts will occur. The mothers' will be assessed at 14 and 36 weeks of pregnancy and at 14 weeks (range 13-15) and 52 (range 48-56) weeks post-delivery. The measurements will be anthropometry, whole body MRI, EchoMRI, and whole body plethysmography (BodPod). The infants' measurements will be anthropometry, whole body MRI, EchoMRI, and whole body plethysmography (PeaPod) for fatness 14 weeks (range 14-15) weeks and 52 (range 48-56) weeks. Mothers and children will have cardio-metabolic risk factors measured in plasma. Data will be collected regarding mothers' dietary intake and physical activity (questionnaires and accelerometry) to assist in counseling. Other data to be collected include questionnaires on quality of life, socio-economic status. Each mother will be followed during pregnancy and for a year post delivery. Each infant will be followed for a year after birth. The researchers have the ability to continue to follow these participants if further funding is forthcoming, as they are all local to the hospital's catchment area and to own physicians.

ELIGIBILITY:
Inclusion Criteria:

* Singleton viable pregnancy
* Gestational age between 9,0 and 15,6
* Body Mass Index of 25 and above
* Age 18 and over
* Ability to contact

Exclusion Criteria:

* Less than 18 years old
* Diagnosis of Diabetes or Hemoglobin A1c (HbA1c)> or = 6.5%
* Known fetal anomaly
* Planned termination of pregnancy
* History of 3 more more consecutive first trimester miscarriages
* Current eating disorder
* Actively suicidal
* Prior or planned bariatric surgery
* Current use of metformin, systemic steroids, antipsychotic agents, anti-seizure medications, mood stabilizers, attention deficit hyperactivity disorder medications
* Continued use of weight loss medication
* Contraindications to aerobic exercise in pregnancy
* Participation in another interventional study that influences weight control
* Enrollment in this trial in a previous pregnancy
* Intention of the participant or of the care provider for the delivery to be outside the Lifestyle Interventions For Expectant (LIFE) Moms consortium hospital
* Participant's unwillingness or inability to commit to a 1 year follow-up of herself or her child, including planning to move away
* Smoking
* History of Drug and/or Alcohol Addiction
* Chronic health problems that prohibit regular exercise or known to influence body composition
* Other chronic disease as determined by investigators
* Claustrophobia (only for participants who elect to have MRI)
* Implanted metal objects that render MRI unsafe (only for participants who elect to have MRI)
* Lack of support from primary health care provider or family members
* Another member of the household is a study participant or staff member
* Any other medical, psychiatric, social or behavioral factor that in the judgement of the Principal Investigator (PI) may interfere with study participation or ability to follow the intervention protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-10; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Infant Percent Fat at Birth | Within 24 hours of birth
  Infant % fat at birth as a continuous variable. This will be ascertained from PeaPod within 24 hours after birth.

SECONDARY OUTCOMES:
Mother fat mass gain 35 Weeks | 35,0-35,6 weeks of pregnancy
  Fat mass gain of mother at 35,0-35,6 weeks of pregnancy as a continuous variable.
Mother fat mass gain one year postpartum | 48-56 weeks postpartum
  Mother's fat mass at 52 (range 48-56) weeks postpartum
Mother's weight one-year postpartum | 48-56 weeks postpartum
  Weight of mother at 52 (range 48-56) weeks
Infant % fat 14 weeks | 13-15 weeks
  Infant %fat at 14 (range 13-15) weeks. This will be ascertained from PeaPod.
Infant % fat 52 weeks | 48-52 weeks
  Infant %fat 52 (range 48-56) weeks.
Infant Weight 14 weeks | 13-15 weeks
  Infant weight at 14 (range 13-15) weeks.
Infant weight 52 weeks | 48-56 weeks
  Infant weight at 52 (range 48-56) weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Dympna Gallagher, EdD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cabre HE, Drews KL, Pomeroy J, Keadle SK, Arteaga SS, Franks PW, Haire-Joshu D, Knowler WC, Pi-Sunyer X, Van Horn L, Wing RR, Cahill AG, Clifton RG, Couch KA, Gallager D, Josefson JL, Joshipura K, Klein S, Martin CK, Peaceman AM, Phelan S, Thom EA, Redman LM; LIFE-Moms Research Group. LIFE-Moms: effects of multicomponent lifestyle randomized control trial on physical activity during pregnancy in women with overweight and obesity. Int J Behav Nutr Phys Act. 2025 Sep 30;22(1):119. doi: 10.1186/s12966-025-01805-9. PMID 41029405
- [Derived] Flanagan EW, Drews KL, Cade WT, Franks PW, Gallagher D, Phelan S, Van Horn L, Redman LM. Metabolic Health and Heterogenous Outcomes of Prenatal Interventions: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2528264. doi: 10.1001/jamanetworkopen.2025.28264. PMID 40839263
- [Derived] Whyte K, Contento I, Wolf R, Guerra L, Martinez E, Pi-Sunyer X, Gallagher D. A secondary analysis of maternal ultra-processed food intake in women with overweight or obesity and associations with gestational weight gain and neonatal body composition outcomes. J Mother Child. 2022 Mar 23;25(4):244-259. doi: 10.34763/jmotherandchild.20212504.d-21-00025. eCollection 2021 Dec 1. PMID 35325513
- [Derived] Redman LM, Drews KL, Klein S, Horn LV, Wing RR, Pi-Sunyer X, Evans M, Joshipura K, Arteaga SS, Cahill AG, Clifton RG, Couch KA, Franks PW, Gallagher D, Haire-Joshu D, Martin CK, Peaceman AM, Phelan S, Thom EA, Yanovski SZ, Knowler WC; LIFE-Moms Research Group. Attenuated early pregnancy weight gain by prenatal lifestyle interventions does not prevent gestational diabetes in the LIFE-Moms consortium. Diabetes Res Clin Pract. 2021 Jan;171:108549. doi: 10.1016/j.diabres.2020.108549. Epub 2020 Nov 22. PMID 33238176
- [Derived] Peaceman AM, Clifton RG, Phelan S, Gallagher D, Evans M, Redman LM, Knowler WC, Joshipura K, Haire-Joshu D, Yanovski SZ, Couch KA, Drews KL, Franks PW, Klein S, Martin CK, Pi-Sunyer X, Thom EA, Van Horn L, Wing RR, Cahill AG; LIFE-Moms Research Group. Lifestyle Interventions Limit Gestational Weight Gain in Women with Overweight or Obesity: LIFE-Moms Prospective Meta-Analysis. Obesity (Silver Spring). 2018 Sep;26(9):1396-1404. doi: 10.1002/oby.22250. Epub 2018 Sep 6. PMID 30230252
- [Derived] Clifton RG, Evans M, Cahill AG, Franks PW, Gallagher D, Phelan S, Pomeroy J, Redman LM, Van Horn L; LIFE-Moms Research Group. Design of lifestyle intervention trials to prevent excessive gestational weight gain in women with overweight or obesity. Obesity (Silver Spring). 2016 Feb;24(2):305-13. doi: 10.1002/oby.21330. Epub 2015 Dec 26. PMID 26708836